CLINICAL TRIAL: NCT05171621
Title: Measuring Subjective Quality of Vision and Metamorphopsia Before and After Epiretinal Membrane and Macular Hole Surgery
Acronym: MQUEST
Status: Completed | Type: Observational
Sponsor: Hayley Westwood (Other)
Responsible Party: Sponsor-Investigator, Hayley Westwood, Senior Clinical Research Officer, University Hospital of Wales
Organization: University Hospital of Wales (Other)
Other Study IDs: 18/NOV/7557
Record Dates: First submitted 2021-11-25; First posted 2021-12-29 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Ophthalmologic Complication; Epiretinal Membrane; Metamorphopsia; Macular Holes
MeSH Terms: conditions — Epiretinal Membrane; Vision Disorders; Retinal Perforations

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Macular holes
- Epiretinal membranes

SUMMARY:
Assessing metamorphopsia and quality of vision pre and post epiretinal and macular hole surgery

DETAILED DESCRIPTION:
Metamorphopsia is a visual symptom in which straight lines appear distorted, for example a vertical window blind may appear wavy which can affect quality of vision. Metamorphopsia is a common symptom in retinal conditions such as epiretinal membranes (ERM) and macular holes. There is a lack of studies analysing the prevalence of ERM in the UK and Europe.

Both of the conditions have shown to be a higher risk factor with age. With an aging population it is likely these numbers will increase. Currently the only treatment option is surgery (vitrectomy) or conservative management to monitor the condition. It would therefore be beneficial to find a tool that would inform the surgeon of a patient's quality of vision and how this impacts their life. A patient's severity of metamorphopsia reveals more precise information on the progression of the disease than visual acuity alone (Nomoto et al. 2013) therefore gaining a better understanding can help aid clinical decisions.

Current clinical practice is to monitor metamorphopsia with an Amsler chart, a grid with lines; the patient is then asked to draw where they can see distortion. They are used to detect metamorphopsia but are unable to quantify and provide an accurate measurement of the severity of metamorphopsia and quality of vision

The Quality of Vision questionnaire (QoV) (McAlinden et al. 2010) is a modern tool developed to specifically measure subjective quality of vision. The Metamorphopsia questionnaire (Arimura et al. 2011) has been developed to provide a measurement of subjective metamorphopsia in macular disease. Both have been psychometrically validated and are in use in a number of clinical trials worldwide.

It would be valuable to investigate the role of each questionnaire in identifying quality of vison and metamorphopsia pre- and post-surgery for ERM and macular holes to establish if there are changes to patient responses. We would compare this to visual acuity and optical coherence tomography (OCT) images pre- and post-surgery to see if changes correspond to the questionnaire responses. If a questionnaire can measure metamorphopsia and its impact on quality of vision in ERM and macular holes, this would assist in clinical decision making.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent
* >18 years old
* Patients listed for epi retinal and macular hole surgery
* Patient is able to perform study procedures

Exclusion Criteria:

* Patients who are diagnosed with a condition other than epiretinal membrane or macular hole

  * Patients not undergoing epiretinal or macular hole surgery
  * Patients will be excluded if there are any complications within surgery, or undergo any procedures that is not an epiretinal or macular hole surgery (i.e vitrectomy, phacoemulsification (lens extraction) as this can affect visual outcomes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have epiretinal membranes or macular holes and have been listed for a vitrectomy
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-10-16 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Compare the responses of the McAllinden and Metamorphopsia Questionnaire | pre surgery and 2 - 3 months post surgery
  analysing changes to responses in the 2 questionnaires pre and post surgery

SECONDARY OUTCOMES:
Changes to BCVA score | Pre surgery and 2-3 months post surgery
  Patients BCVA pre and post surgery to see if there is an improvement

OTHER OUTCOMES:
Assess correlations between the Mcallinden and Metamorphopsia questionnaire scores and objective clinical parameters | Pre surgery and 2-3 month post surgery
  do the questionnaires show changes pre and post surgery and do they match clinical outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Wales, Cardiff, United Kingdom

IPD SHARING:
Plan to Share IPD: No